CLINICAL TRIAL: NCT00937560
Title: A Single-arm Phase II Clinical Study Investigating the Addition of Bevacizumab to Carboplatin and Weekly Paclitaxel as First-line Treatment in Patients With Epithelial Ovarian Cancer
Brief Title: A Study of First Line Treatment With Avastin (Bevacizumab) in Combination With Carboplatin and Weekly Paclitaxel in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO22225; 2008-008336-85 (EudraCT Number)
Record Dates: First submitted 2009-07-06; First posted 2009-07-13 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Paclitaxel; Carboplatin

ARMS (1):
- Bevacizumab + paclitaxel + carboplatin (Experimental): Participants received 6-8 (at the investigator's discretion) 3-week cycles of bevacizumab 7.5 mg/kg intravenously (iv) on Day 1 of each cycle, paclitaxel 80 mg/m^2 iv on Days 1, 8, and 15 of each cycle, and carboplatin iv to an area under the curve of 6 on Day 1 of each cycle. The initial dose of carboplatin was calculated according to the Calvert formula (mg = [glomerular filtration rate + 25] x 6). Following the combination treatments, participants received up to 17 3-week cycles of bevacizumab 7.5 mg/g iv alone.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was supplied as a sterile solution for infusion.
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel was supplied locally in commercial batches.
  Other Names: Taxol
Drug: Carboplatin — Carboplatin was supplied locally in commercial batches.
  Other Names: Paraplatin

SUMMARY:
This single arm study evaluated the efficacy and safety of first-line chemotherapy with carboplatin and dose-dense weekly paclitaxel plus bevacizumab (Avastin) in participants with epithelial ovarian, fallopian tube, or primary peritoneal cancer. Participants received 6-8 3-week cycles of treatment with bevacizumab 7.5 mg/kg intravenously (iv) on Day 1 of each cycle, paclitaxel 80 mg/m^2 iv on days 1, 8, and 15 of each cycle, and carboplatin iv to an area under the curve (AUC) of 6 on day 1 of each cycle. Following combination chemotherapy, bevacizumab could be continued to be given as a monotherapy.

ELIGIBILITY:
Inclusion Criteria

* Female patients, ≥ 18 years of age.
* Epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Initial surgery, but no chemotherapy or radiotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria

* Non-epithelial tumors.
* Ovarian tumors with low malignant potential.
* Previous systemic anti-cancer therapy for ovarian cancer.
* History or evidence of synchronous primary endometrial cancer.
* Current or recent daily treatment with aspirin (> 325mg/day) or with full dose anticoagulant or thrombolytic agents for therapeutic purposes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-06-25 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2013-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (55):
- Brazil (2):
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clinicas - FMUSP, Oncologia, São Paulo, São Paulo
- France (18):
  - Centre Hospitalier Henri Duffaut; Hematologie, Avignon
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Ch De Brive La Gaillarde; Radiotherapie Oncologie, Brive-la-Gaillarde
  - Hopital Antoine Beclere; Service de Medecine Interne, Clamart
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Chi Alpes Du Sud Site De Gap; Med Interne Et Polyvalente, Gap
  - Institut Daniel Hollard, Grenoble
  - Hôpital Saint Joseph; Oncologie Medicale, Marseille
  - CHRA;Hematologie, Metz-Tessy
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - GH Paris Saint Joseph; Hopital De Jour Oncologie, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Hopital De La Miletrie; Hematologie Et Oncologie Medicale, Poitiers
  - Institut de Cancerologie de La Loire; Radiotherapie, Saint-Priest-en-Jarez
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
- Italy (4):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica B, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - Universita' Cattolica Del Sacro Cuore; Reparto Ginecologia Oncologica, Rome, Lazio
  - Universita' Cattolica Del Sacro Cuore; Reparto Ginecologia Oncologica, Campobasso, Molise
- Netherlands (7):
  - Medisch Centrum Alkmaar, Alkmaar
  - Academisch Medisch Centrum; Inwendige Geneeskunde, Amsterdam
  - Medisch Spectrum Twente Enschede; Internal Medicine, Enschede
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Mc Haaglanden, Locatie Antoniushove; Interne Geneeskunde, Leidschendam
  - Sint Elizabeth Ziekenhuis; Inwendige Geneeskunde, Tilburg
  - Isala Klinieken, Locatie Sophia; Inwendige Geneeskunde, Zwolle
- Norway (2):
  - The Norvegian Radium Hospital Montebello; Dept of Oncology, Oslo
  - St. Olavs Hospital; Kvinneklinikken, Trondheim
- Russia (7):
  - Regional Clinical Oncology Dispensary, Krasnodar
  - Oncology Hospital; Chemotherapy Dept., Moscow
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow
  - City Clinical Oncology Hospital, Moscow
  - Medical Radiological Scientific Center; Department of Radiotherapy of Gynaecological Disease, Obninsk, Kaluzhskaya Region
  - St. Petersburg Oncology & Gynecology; City Clinical Oncology Dispensary, Saint Petersburg
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
- Spain (9):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset; Onkology, Gothenburg
  - Uni Hospital Linkoeping; Dept. of Oncology, Linköping
  - Örebro University Hospital; Department of Gynecologic Oncology, Örebro
  - Norrlands Uni Hospital; Onkologi Avd., Umeå
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Royal Marsden Hospital; Dept of Med-Onc, London, United Kingdom

REFERENCES:
- [Derived] Gonzalez-Martin A, Gladieff L, Tholander B, Stroyakovsky D, Gore M, Scambia G, Kovalenko N, Oaknin A, Ronco JP, Freudensprung U, Pignata S; OCTAVIA Investigators. Efficacy and safety results from OCTAVIA, a single-arm phase II study evaluating front-line bevacizumab, carboplatin and weekly paclitaxel for ovarian cancer. Eur J Cancer. 2013 Dec;49(18):3831-8. doi: 10.1016/j.ejca.2013.08.002. Epub 2013 Sep 2. PMID 24007819

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Paclitaxel + Carboplatin: Participants received 6-8 (at the investigator's discretion) 3-week cycles of bevacizumab 7.5 milligrams per kilograms (mg/kg) intravenously (IV) on Day 1 of each cycle, paclitaxel 80 milligrams per square meters of body surface (mg/m^2) IV on Days 1, 8, and 15 of each cycle, and carboplatin IV to an area under the curve (AUC) of 6 on Day 1 of each cycle. The initial dose of carboplatin was calculated according to the Calvert formula (milligrams [mg] equals [=] [glomerular filtration rate (GFR) + 25] x 6). Following the initial treatment (bevacizumab + paclitaxel + carboplatin) period, participants received additional 3-week cycles of monotherapy bevacizumab 7.5 mg/kg IV during the maintenance treatment period. The total maximum bevacizumab treatment duration was 17 cycles, (12 months) which included both the initial treatment period and the bevacizumab monotherapy maintenance treatment period.
Period: Initial Treatment
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Started | 189
Received Treatment | 189
Completed | 168
Not Completed | 21
Not completed — Death | 6
Not completed — Withdraw consent | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — No end of study page | 10
Period: Maintenance Treatment
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Started | 168
Completed | 150
Not Completed | 18
Not completed — Death | 12
Not completed — Withdraw consent | 5
Not completed — According to protocol | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All enrolled participants who received at least 1 dose of any study medication (bevacizumab, carboplatin or paclitaxel).
Groups:
- Bevacizumab + Paclitaxel + Carboplatin: Participants received 6-8 (at the investigator's discretion) 3-week cycles of bevacizumab 7.5 mg/kg IV on Day 1 of each cycle, paclitaxel 80 mg/m^2 IV on Days 1, 8, and 15 of each cycle, and carboplatin IV to an AUC of 6 on Day 1 of each cycle. The initial dose of carboplatin was calculated according to the Calvert formula (mg = [GFR + 25] x 6). Following the initial treatment (bevacizumab + paclitaxel + carboplatin) period, participants received additional 3-week cycles of monotherapy bevacizumab 7.5 mg/kg IV during the maintenance treatment period. The total maximum bevacizumab treatment duration was 17 cycles, (12 months) which included both the initial treatment period and the bevacizumab monotherapy maintenance treatment period.
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 189
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first administration of any study treatment to the first disease progression using Response Evaluation Criteria In Solid Tumors (RECIST) or death from any cause, whichever occurred first.
Time Frame: Baseline to the data cut-off date of 19 Jul 2012 for analysis of the primary Outcome Measure (follow-up time up to 3 years, 1 month)
Population: Intent-to-treat population: All enrolled participants who received at least 1 dose of any study medication (bevacizumab, carboplatin, or paclitaxel).
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 189
Months | 23.7 [19.9 to 26.4]

2. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as either a complete response (CR) or a partial response (PR). Using the Response Evaluation Criteria in Solid Tumors (RECIST), a CR was defined as the disappearance of all target lesions and all non-target lesions, normalization of tumor marker level, and no new lesions and a PR was defined as the disappearance of all target lesions and persistence of ≥ 1 non-target lesions and/or the maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diameter of target lesions, and no new lesions or unequivocal progression of existing non-target lesions. Only participants with measurable disease were included in the analysis according to RECIST only. Only participants with a Baseline ovarian cancer mucin CA-125 level ≥ 2 times the upper limit of normal who had a ≥ 50% reduction of CA-125 from Baseline were included in the analysis according to CA-125 level.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 126
Percentage of participants
  RECIST only (N=91) | 84.6 [75.5 to 91.3]
  CA-125 level only (N=101) | 97.0 [91.6 to 99.4]
  RECIST and CA-125 level combined (N=126) | 92.1 [85.9 to 96.1]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the interval between the date of the first documented response by RECIST to the date of first disease progression or death, whichever occurred earlier. Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of 1 or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Only participants with measurable disease were included in the analysis according to RECIST only. Only participants with a Baseline ovarian cancer mucin CA-125 level ≥ 2 times the upper limit of normal who had a ≥ 50% reduction of CA-125 from Baseline were included in the analysis according to CA-125 level.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 116
Months
  RECIST only (N=77) | 14.7 [12.7 to 16.1]
  CA-125 level only (N=98) | 17.5 [15.4 to 21.9]
  RECIST and CA-125 level combined (N=116) | 17.4 [15.4 to 21.9]

4. Secondary Outcome: Overall Survival at 1 Year and 2 Years
Description: Reported are the percentage of participants that were alive at 1 year and 2 years after enrolling in the study.
Time Frame: Baseline to Year 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 189
Percentage of participants
  Year 1 | 97.7 [95.4 to 99.9]
  Year 2 | 92.1 [88.0 to 96.2]

5. Secondary Outcome: Biological Progression-free Interval
Description: Biological progression-free interval is defined as the interval from the date of the first administration of any study treatment to the date of the first documented serial elevation of the ovarian cancer mucin CA-125. More precisely, this is defined as the first documented increase in CA-125 levels as follows: (1) CA-125 greater than or equal to 2 times the upper level of normal (ULN) on 2 occasions at least 1 week apart (for patients with CA-125 within normal range pre-treatment) or (2) CA-125 greater than or equal to 2 times the ULN on 2 occasions at least 1 week apart (for patients with elevated CA-125 pre-treatment and initial normalisation of CA-125 on-treatment) or (3) CA-125 greater than or equal to 2 times the nadir value, which is the lowest observed CA-125 value per patient on 2 occasions at least 1 week apart (for patients with elevated CA-125 pre-treatment which never normalised).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 189
Months | NA [NA to NA] — The median and the limits of the 95% confidence interval could not be calculated due to too few events.

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (up to 4 years, 1 month)
Description: Safety population: All enrolled participants who received at least 1 dose of any study medication (bevacizumab, carboplatin, or paclitaxel).
Groups:
- Bevacizumab + Paclitaxel + Carboplatin: Participants received 6-8 (at the investigator's discretion) 3-week cycles of bevacizumab 7.5 mg/kg intravenously (iv) on Day 1 of each cycle, paclitaxel 80 mg/m^2 iv on Days 1, 8, and 15 of each cycle, and carboplatin iv to an area under the curve of 6 on Day 1 of each cycle. The initial dose of carboplatin was calculated according to the Calvert formula (mg = [glomerular filtration rate + 25] x 6). Following the combination treatments, participants received up to 17 3-week cycles of bevacizumab 7.5 mg/g iv alone. Bevacizumab: Bevacizumab was supplied as a sterile solution for infusion. Paclitaxel: Paclitaxel was supplied locally in commercial batches. Carboplatin: Carboplatin was supplied locally in commercial batches.
Arm/Group | Bevacizumab + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 43/189
Other Adverse Events (participants affected / at risk) | 186/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Carboplatin (N=189)
Subileus (Gastrointestinal disorders) | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Oesophagits (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Infected lymphocele (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism venous (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Pyrexia (General disorders) | 2
Chest discomfort (General disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Carboplatin (N=189)
Neutropenia (Blood and lymphatic system disorders) | 153
Thrombocytopenia (Blood and lymphatic system disorders) | 85
Anaemia (Blood and lymphatic system disorders) | 111
Leukopenia (Blood and lymphatic system disorders) | 48
Lymphopenia (Blood and lymphatic system disorders) | 14
Thrombocytosis (Blood and lymphatic system disorders) | 11
Nausea (Gastrointestinal disorders) | 87
Diarrhoea (Gastrointestinal disorders) | 59
Constipation (Gastrointestinal disorders) | 64
Stomatitis (Gastrointestinal disorders) | 39
Vomiting (Gastrointestinal disorders) | 43
Abdominal pain (Gastrointestinal disorders) | 31
Abdominal pain upper (Gastrointestinal disorders) | 20
Gingival bleeding (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 105
Asthenia (General disorders) | 22
Pyrexia (General disorders) | 19
Mucosal inflammation (General disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 80
Headache (Nervous system disorders) | 34
Paraesthesia (Nervous system disorders) | 25
Dysgeusia (Nervous system disorders) | 22
Dizziness (Nervous system disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 89
Rash (Skin and subcutaneous tissue disorders) | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 15
Erythema (Skin and subcutaneous tissue disorders) | 10
Nail toxicity (Skin and subcutaneous tissue disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 19
Hypokalaemia (Metabolism and nutrition disorders) | 16
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 76
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Urinary tract infection (Infections and infestations) | 21
Upper respiratory tract infection (Infections and infestations) | 18
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 17
Hypertension (Vascular disorders) | 44
Alanine aminotransferase increased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 14
Proteinuria (Renal and urinary disorders) | 11
Insomnia (Psychiatric disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.